CLINICAL TRIAL: NCT06376747
Title: The Influence of Blood Sampling Technique on the Total Amount of Blood Collected for Laboratory Testing in Critically Ill Pediatric Patients: a Prospective Randomized Study
Brief Title: The Influence of Blood Sampling Technique on the Total Amount of Blood Collected for Laboratory Testing Critically Ill Pediatric Patients
Acronym: PEDPBM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, prof. Petr Stourac M.D., Ph.D., MBA, FESAIC, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: KDAR- PBM 2024
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Iatrogenic Anaemia
Keywords: Paediatric patient; Patient Blood Management; Paediatric ICU

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Patients will be randomized into two groups: a group with standard blood sampling technique and a group with closed technique blood sampling by using randomizing software.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard blood sampling technique (Active Comparator): Blood withdrawal after catheter decontamination, blood draw for laboratory analysis, catheter flush
  Interventions: Procedure: Standard blood sampling technique
- Closed technique blood sampling (Experimental): In-line sampling: through 2 three-way stopcocks: blood withdrawal for catheter decontamination, blood draw for laboratory analysis, return of the withdrawn blood for catheter decontamination, catheter flush
  Interventions: Procedure: In line sampling

INTERVENTIONS:
Procedure: In line sampling — closed technique of sample collection
  Arms: Closed technique blood sampling
Procedure: Standard blood sampling technique — Blood draws using standard steps: blood withdrawal for catheter, decontamination (disposed),blood draw for laboratory analysis,catheter flush
  Arms: Standard blood sampling technique

SUMMARY:
The aim of this prospective randomized study is to evaluate blood loss caused by laboratory blood draws in patients in the paediatric ICU (Intensive Care Unit) of a tertiary hospital among two groups of patients with established long-term or mid-term intravenous access. In the first group, patients will undergo blood draws using the standard method. In the second group of patients, blood draws will be performed using a closed system.

DETAILED DESCRIPTION:
Anaemia is one of the most common comorbidities among patients hospitalized in intensive care units. Hospital-acquired anaemia (HAA) is a newly developed anaemia that occurs during hospitalization in patients who were not anaemic prior to admission. Patients with HAA have a higher risk of developing complications such as infections, muscle weakness, and neurocognitive developmental disorders; an increased incidence of blood and blood product transfusions (and related complications); longer hospital stays, and higher morbidity and mortality. According to available data, the incidence of anaemia in adults hospitalized in the ICU ranges from 40 to 74%. There a feq data describing anemia in critically ill pediatric patients, with the estimated incidence being up to 50%.

The etiology of HAA is multifactorial and is related to the severity of the underlying disease (sepsis, coagulation disorders, bleeding, renal failure, malnutrition, bone marrow suppression, decreased erythropoietin production, etc.). Another factor contributing to the development of anaemia in critically ill patients is iatrogenic blood loss caused by blood draws for laboratory testing.

In addition to the standard blood collection method, closed-loop sampling (in-line sampling) can also be used, with studies in adult patients showing a reduction in the amount of blood drawn, ranging from 20 to 80% after its implementation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for the study.
* Patients with established intravenous access: CVC (Central Venous Catheter), CICC (Centrally Inserted Central Catheter), PICC (Peripherally Inserted Central Catheter), MVC (Midline Venous Catheter), venous port, from which blood can be drawn.
* Anticipated length of stay in the ICU more than 24 hours

Exclusion Criteria:

* Age outside the specified range.
* Peripheral venous access only.
* Anticipated length of stay in the ICU less than 24 hours.
* Organ donors.
* Lack of consent from the legal representative/patient.

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Average amount of blood collected for laboratory diagnostic purposes | On day 1,3,5,7,10,14 and 28 of patient stay at paediatric ICU
  Average amount of blood collected for laboratory diagnostic purposes on days 1, 3, 5, 7, 10, 14, and 28 of hospitalization in two groups of patients subjected to different blood sampling techniques for laboratory testing

SECONDARY OUTCOMES:
Cumulative amount of blood drawn per day of ICU hospitalization | On the day of patient' s discharge from paediatric ICU
  Cumulative amount of blood drawn, relative to the patient's body weight and age, per day of ICU hospitalization
Absolute amount of blood drawn and blood used for laboratory testing | On the day of patient' s discharge from paediatric ICU
  Absolute amount of blood drawn and blood used for laboratory testing, relative to the patient's body weight, age, and day of ICU hospitalization
Trend of haemoglobin decline over time | Ondays 1,3,5,7,10,14 and 28 of patient stay at paediatric ICU
  Trend of haemoglobin decline over time, defined as the absolute value of haemoglobin
Incidence of anaemia | on the day of patient' s discharge from paediatric ICU
  decrease in haemoglobin levels below 90 g/l at any time during hospitalization
Incidence of anaemia up to transfusion trigger | on the day of patient' s discharge from paediatric ICU
  haemoglobin levels below 70 g/l at any time during hospitalization
Frequency of blood product transfusions and their quantity | on the day of patient' s discharge from paediatric ICU
  Frequency of blood product transfusions (erythrocytes, platelets, plasma, fibrinogen, and other coagulation factors) and their quantity relative to the patient's body weight and age
Type and frequency of laboratory tests | on the day of patient' s discharge from paediatric ICU
  Type and frequency of laboratory tests noted on daily basis by ICU nursing stuff
Incidence of coagulopathy | on the day of patient' s discharge from paediatric ICU
  Incidence of coagulopathy defined as INR above 1.4 and/or aPTT above 1.5 and/or fibrinogen below 1.5 g/l
Incidence of catheter-related complications | on the day of patient' s discharge from paediatric ICU
  Incidence of catheter-related complications catheter infections, catheter occlusion defined, accidental catheter withdrawal)
Time to catheter replacement in case of catheter exchange | on the day of patient' s discharge from paediatric ICU
  Time to catheter replacement in case of catheter exchange (in days)

CONTACTS AND LOCATIONS:
Locations (1):
- KDAR - department of pediatrics anesthesia and resuscitation, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided